CLINICAL TRIAL: NCT04303481
Title: The Effect of Consuming Enzymes and Prebiotics on Body Composition and Blood Biochemical Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-062-A
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Gut Microbiota
Keywords: Anthropometric index; Biochemical items

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal diet (Other)
  Interventions: Other: normal diet
- weight loss program kit (Experimental)
  Interventions: Other: weight loss program kit
- weight loss program kit with A. muciniphila prebiotics (Experimental)
  Interventions: Other: weight loss program kit with A. muciniphila prebiotics

INTERVENTIONS:
Other: normal diet — Control
  Arms: normal diet
Other: weight loss program kit — Subjects should adhere to the eating plan, which contained the following kit components : four flavors of collagen drinks [i.e., Caviar Collagen Enzyme Drink, Collagen Enzyme Drinks (Peach Taste), Collagen Enzyme Drinks (Grape Fruit Taste), Saussurea involucrata Enzyme Drink (Litchi Taste)], six flavors of mike shakes (i.e., Corn Soup Mike Shake, Strawberry Mike Shake, Chocolate Mike Shake, Vanilla Mike Shake, Banana Mike Shakes, Matcha Mike Shakes), Fruit and Vegitable Congee, and Botanical Liquid Sachet.
  Arms: weight loss program kit
Other: weight loss program kit with A. muciniphila prebiotics — Subjects should adhere to the eating plan, which contained the following kit components : four flavors of collagen drinks [i.e., Caviar Collagen Enzyme Drink, Collagen Enzyme Drinks (Peach Taste), Collagen Enzyme Drinks (Grape Fruit Taste), Saussurea involucrata Enzyme Drink (Litchi Taste)], six flavors of mike shakes (i.e., Corn Soup Mike Shake, Strawberry Mike Shake, Chocolate Mike Shake, Vanilla Mike Shake, Banana Mike Shakes, Matcha Mike Shakes), Fruit and Vegitable Congee, Botanical Liquid Sachet, and Probiotics Liquid Sachet
  Arms: weight loss program kit with A. muciniphila prebiotics

SUMMARY:
To assess the effects of consuming enzymes and prebiotics on improvement of weight loss and biochemical parameters

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 20 and 50 years old
* Body mass index (BMI) ≥ 22 (kg/m^2) or body fat mass: male > 25%, female > 30%
* Prohibitions on other nutritional supplements (probiotics and prebiotics) before two weeks of the study
* Abidance by the similar diet and exercise habits over the study.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Menopausal woman
* Diabetes mellitus
* Implementation in weight loss programs before a half year of this study
* Metabolic disorders
* Kidney diseases
* Liver diseases
* Cardiovascular diseases
* Nervous system diseases
* Gastrointestinal diseases
* Heavy drinking or constant drug use.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change of body fat mass | Months 0, 1 and 2
  The body fat mass (kg) was assessed by InBody770.
The change of Triglyceride | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of Triglyceride
The change of Total cholestrol | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of Total cholestrol
The change of HDL-cholestrol | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of HDL-cholestrol
The change of LDL-cholestrol | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of LDL-cholestrol
Fecal microbiome analysis | Months 0, 1 and 2
  Firmicutes, Bacteroidetes, Lactobucillius, and A. muciniphila were quantified by quantitative PCR.
The change of body mass index (BMI) | Months 0, 1 and 2
  BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass.The body mass index (BMI, kg/m^2) and body mass (kg) were assessed by InBody770.
The change of body fat percentage | Months 0, 1 and 2
  The body fat percentage (%) was assessed by InBody770.
The change of visceral fat | Months 0, 1 and 2
  The visceral fat (10 cm^2) was assessed by InBody770.

SECONDARY OUTCOMES:
The change of fasting glycemia | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of fasting glycemia
The change of aspartate aminotransferase | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of aspartate aminotransferase
The change of alanine aminotransferase | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of alanine aminotransferase
The change of albumin | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of albumin
The change of creatine | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of creatine
The change of uric acid | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of uric acid
The change of white blood cell | Months 0, 1 and 2
  Venous blood was sampled to measure concentrations of white blood cell

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Han Wu, Principal Investigator — Study Principal Investigator
Locations (1):
- National Pingtung University of Science and Technology, Pingtung City, Neipu Township, Taiwan